CLINICAL TRIAL: NCT01914471
Title: A Community-Academic Partnership to Address Disparities in Obesity Among Youth
Brief Title: A Randomized Controlled Trial of Students for Nutrition and eXercise
Acronym: SNaX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R24MD001648 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): These schools did not receive the intervention.
- Students for Nutrition and eXercise (Experimental): These schools received the entirety of Students for Nutrition and eXercise, a middle-school-based obesity-prevention intervention combining school-wide environmental changes, multimedia, encouragement to eat healthy school cafeteria foods, and peer-led education and marketing
  Interventions: Behavioral: Students for Nutrition and eXercise

INTERVENTIONS:
Behavioral: Students for Nutrition and eXercise — These schools received the entirety of Students for Nutrition and eXercise, a middle-school-based obesity-prevention intervention combining school-wide environmental changes, multimedia, encouragement to eat healthy school cafeteria foods, and peer-led education and marketing
  Arms: Students for Nutrition and eXercise

SUMMARY:
Objectives: We conducted a randomized controlled trial (RCT) of Students for Nutrition and eXercise (SNaX), a middle-school-based obesity-prevention intervention combining school-wide environmental changes, multimedia, encouragement to eat healthy school cafeteria foods, and peer-led education and marketing.

Methods: We randomly selected schools from the Los Angeles Unified School District (LAUSD) and assigned five to the intervention group and five to a wait-list control group. School records were obtained for number of fruits and vegetables served, students served lunch, and snacks sold per attending student. Pre- and post-intervention surveys assessed psychosocial variables among 2,997 seventh-graders (75% of all seventh-graders across schools).

Hypotheses: For the RCT of SNaX, we hypothesized that SNaX would lead to increases in the proportion of students served in the cafeteria (because SNaX markets cafeterias' healthy foods); increased fruit and vegetable servings (because SNaX increases access to sliced/bite-sized fruits and vegetables); decreased school store snack sales; and greater water consumption. We also hypothesized that SNaX would lead to more positive attitudes about the cafeteria and water, improve obesity-prevention knowledge, and increase intentions to drink water.

ELIGIBILITY:
Inclusion Criteria:

* schools with >50% NSLP-eligible students (a proxy for low-income) and <900 - seventh-graders

Exclusion Criteria:

* schools with <50% NSLP-eligible students and >900 seventh-graders

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2997 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of students obtaining lunch per day by National School Lunch Program (NSLP) eligibility | 5 months
  We obtained the number of students obtaining lunch per day (by National School Lunch Program (NSLP) eligibility) from schools.
Number of fruits and vegetables served per day | 5 months
  We obtained the number of fruits and vegetables served per day from the school cafeterias.

SECONDARY OUTCOMES:
Attitudes about the cafeteria | 5 months
  Attitudes about the cafeteria were calculated by survey data using the mean of two 7-point scales representing attitudes about the cafeteria: unsatisfying/satisfying and bad for my health/good for my health.
Attitudes about water | 5 months
  Attitudes about water were measured with a survey including an 11-point scale (very negatively/very positively).
Knowledge about healthy eating and physical activity | 5 months
  Knowledge about healthy eating and physical activity was measured with a survey containing 6 true/false items.
Intentions to drink water | 5 months
  Intentions to drink water were assessed with two survey items, "How likely is it that you will drink water [or drink water from a refillable water bottle] the next day you are in school?" with 5-point scales (extremely likely/extremely unlikely).
Water consumption frequency | 5 months
  Water consumption frequency was assessed by survey with, "How often do you usually drink tap water?" and "How often do you usually use a refillable water bottle to drink water?" (every day, a few times a week, once a week, twice a month, once a month, less than once a month, never).
Number of snacks sold per day | 5 months
  We obtained the data on the number of snacks sold per day from the school store.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Schuster, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- RAND Corporation, Santa Monica, California, United States

REFERENCES:
- [Derived] Bogart LM, Cowgill BO, Elliott MN, Klein DJ, Hawes-Dawson J, Uyeda K, Elijah J, Binkle DG, Schuster MA. A randomized controlled trial of students for nutrition and eXercise: a community-based participatory research study. J Adolesc Health. 2014 Sep;55(3):415-22. doi: 10.1016/j.jadohealth.2014.03.003. Epub 2014 Apr 29. PMID 24784545